CLINICAL TRIAL: NCT04899401
Title: A Randomized, Open, Controlled Study to Evaluate the Efficacy and Safety of PediaFlù® (Dietary Supplement) Along With Standard of Care in Children With Acute Tonsillopharyngitis / Rhinopharyngitis Versus Standard of Care Only
Brief Title: Trial To Assess Efficacy and Safety of PediaFlu® in Children With Acute Tonsillopharyngitis / Rhinopharyngitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatrica S.r.l (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPPED/0120/FS
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-06

CONDITIONS: Tonsillopharyngitis; Rhinopharyngitis
Keywords: ATP; tonsillopharyngitis; Rhinopharyngitis; PediaFlù®; Pelargonium sidoides; Propolis
MeSH Terms: conditions — Nasopharyngitis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, multicenter clinical investigation, with two parallel groups of subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care +PediaFlù® (Experimental)
  Interventions: Dietary Supplement: Standard of care + PediaFlù®
- Standard of care (Active Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Dietary Supplement: Standard of care + PediaFlù® — Standard of care: Standard of care for acute tonsillitis / rhinopharyngitis is focused on symptomatic treatment. PediaFlù®: During the 6 days of the clinical investigation, the subjects will administer PediaFlù® 5ml x3 times per day for children below 6 years and 10mlx3 times per day for children above 6 years.
  Arms: Standard of care +PediaFlù®
Other: Standard of care — Standard of care for acute tonsillitis / rhinopharyngitis is focused on symptomatic treatment. Standard of care Nasopharyngeal liberation through hydration with drinking fluids to support body fluid excretion, aspiration of secretions, NaCl solution for nasal irrigation, Nasal sprays with sea water, nasal spray with active compound (to be used only at special indication of the medical doctor) Throat spray with Benzydamine hydrochloride (Tantum Verde®), Pediatric use: children over 6 and below 12: 4 sprays 2 - 6 times a day. Children (under 6 years): 1 spray per 4 kg of body weight, a maximum of 4 sprays at once, 2-6 times a day according to the leaflet. Each spray equals 0.17 ml of solution. Acetaminophen (Paracetamol) per os: at need, as antipyretic (>38,5C), 10 mg/kg/dose, per need every 6-8 hours or according to the leaflet, maximum dosage 80 mg / kg / day. A dosage of over 30 mg/Kg/dose will result in an IP failure;
  Arms: Standard of care

SUMMARY:
Sore throat or acute tonsillopharyngitis, often referred to as angina catarrhalis in Central and Eastern Europe, affects mainly children, adolescents and young adults and represents one of the most common reasons to consult a family physician. While most patients complaining of sore throats have an infection, it has been estimated that fewer than 20% present with a clear indication for antibiotic therapy, i.e., are positive for hemolytic streptococcus.

Acute tonsillopharyngitis (ATP) is a highly prevalent, seasonal infective disorder characterized by an inflammation of the pharynx and the palatine tonsils, which occurs in all age groups and accounts for about 5% of all visits in pediatric care. Common symptoms of ATP include sore throat, dysphagia, red pharynx, enlarged tonsils sometimes covered with exudate, fever with sudden onset, malaise, gastrointestinal complaints, halitosis, rhinorrhea and cough. Children with non-streptococcal tonsillopharyngitis are often over-treated with antibiotics.

The scientific literature currently available shows that the extract of Pelargonium sidoides may be effective in the treatment of disorders affecting the respiratory tract.

Evidence shows that zinc is beneficial for the common cold in healthy children and adults living in high-income countries and it may inhibit replication of the virus. In addition, zinc (lozenges or syrup) reduces the average duration of the common cold in healthy people assuming zinc within 24 hours of onset of symptoms Propolis has been widely investigated for its antibacterial, antiviral, and anti-inflammatory properties and is administered as an add-on therapy during watchful waiting for better control of symptoms in non-streptococcal pharyngitis.

The above-mentioned considerations, have suggested Pediatrica Srl to develop a food supplement specific for pediatric age for the well-being of the airways (PediaFlù®). This product is actually on the market as adjuvant in seasonal diseases.

The present clinical investigation is planned to verify and confirm these encouraging results in a setting of standard clinical practice.

This is a randomized, open, controlled study to evaluate the efficacy and safety of PediaFlù® (dietary supplement) along with standard of care in children with acute tonsillopharyngitis / rhinopharyngitis versus standard of care only.

The primary objective is to evaluate the efficacy and safety of the tested dietary supplement administered along with standard care vs standard care alone in children affected by acute tonsillopharyngitis (ATP).

The secondary objectives of the study are the assessment of the use of rescue medicine (Ibuprofen or high dose of Paracetamol) and the evaluation of the overall improvement symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion if all the following criteria are respected:
* male and female (children 3 - 10 years old);
* acute tonsillitis / rhinopharyngitis (sore throat, catarrhal angina), duration of complaints ≤ 48 hours,
* Absence of pharyngeal exudate and/or Mc Isaac score 0-1 + negative rapid test for β-hemolytic streptococcus and SARS-CoV-2 identification
* tonsillitis symptoms score (TSS) ≥ 8 points,
* both parents capable of and freely willing to provide written informed consent prior to participating in the clinical investigation.
* for children above 6 years old capable willing to provide written informed consent prior to participating in the clinical investigation.

Exclusion Criteria:

* evidence of lacunar or follicular angina.
* more than two episodes of tonsillitis within the last 12 months,
* mandatory indication for therapy with antibiotics (e.g., abscess, septic tonsillitis, history of rheumatic fever, post-streptococcus glomerulonephritis, and chorea minor Sydenham),
* history of close contact with SARS-COV-2 infected individuals in the last 10 days before symptoms onset
* treatment with antibiotics within 4 months prior to study inclusion,
* increased hemorrhagic diathesis, chronic diseases (e.g. severe heart, kidney or liver diseases), immunosuppression,
* known or suspected hypersensitivity to study medication,
* concomitant treatment potentially influencing study outcome or known interactions with study medication (e.g., coumarin derivatives),
* participation in another clinical study within the last 3 months prior to clinical investigation inclusion.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Tonsillitis severity score | 6 days
  Tonsillitis severity score (TSS) Intensity score in between 0 and 3. The results will be compared in terms of absolute change of tonsillitis severity score from baseline to final visit, between groups and intra-groups;
Number of treatment failure | 6 days
  The result of using rescue medicine (Ibuprofen or dosage of over 30 mg/Kg/dose daily of paracetamol) will be compared in the two groups.
AE/SAE incidence. | 6 days
  Adverse Events/Serious Adverse Events incidence.

SECONDARY OUTCOMES:
Compliance | 6 days
  IP compliance (the amount of IP ingested divided by the value the subject should have ingested and multiplied by 100);
Symptoms improvement | 6 days
  Overall symptoms improvement through IGAE (Investigator Global Assessment of Efficacy), a 4-point scale: 1= very good efficacy, 2 = good efficacy, 3 = moderate efficacy and 4 = poor efficacy.

CONTACTS AND LOCATIONS:
Locations (3):
- Romania (3):
  - CMMF Dr. Morariu Bordea Maria, Timișoara, Timiș County
  - CM Dr. Herteg Dorina, Timișoara, Timiș County
  - CM Dr. Matei Cristian-Radu, Timișoara

REFERENCES:
- [Derived] Cardinale F, Barattini DF, Centi A, Giuntini G, Bordea MM, Herteg D, Barattini L, Matei CR. Open, Randomised, Controlled Study to Evaluate the Role of a Dietary Supplement Containing Pelargonium sidoides Extract, Honey, Propolis, and Zinc as Adjuvant Treatment in Children with Acute Tonsillopharyngitis. Children (Basel). 2025 Mar 10;12(3):345. doi: 10.3390/children12030345. PMID 40150627
- [Derived] Cardinale F, Barattini DF, Sbrocca F, Centi A, Giuntini G, Morariu Bordea M, Herteg D, Rosu S, Matei CR. The Effects of a Dietary Supplement (PediaFlu) Plus Standard of Care in Children With Acute Tonsillopharyngitis/Rhinopharyngitis: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 May 31;13:e53703. doi: 10.2196/53703. PMID 38819917